CLINICAL TRIAL: NCT00607477
Title: A Pilot Study of the Treatment of VEGF-Signaling Pathway Inhibitor-Induced Hypertension With Direct Vasodilators, Minoxidil and Hydralazine
Brief Title: Pilot Study of the Treatment of Vascular Endothelial Growth Factor(VEGF)Signaling Pathway Inhibitor-Induced Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been terminated due to poor accrual.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15386B
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Treatment Induced Hypertension
MeSH Terms: interventions — Minoxidil; Hydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Minoxidil
  Interventions: Drug: Minoxidil
- 2 (Active Comparator): Hydralazine
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Minoxidil — 2.5 mg taken twice daily for 1 week, followed by 5 mg taken twice daily for the next week, followed by 10 mg twice daily for the next week
  Arms: 1
Drug: Hydralazine — 25 mg taken twice daily for 1 week, followed by 50 mg taken twice daily for the next week, followed by 100 mg twice daily for the next week
  Arms: 2

SUMMARY:
The purpose of this study is to describe the length of time and extent of blood pressure response to minoxidil and hydralazine among cancer patients with difficult-to-treat vascular endothelial growth factor (VEGF) inhibitor treatment induced hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing treatment for malignancy by at the University of Chicago with any agent with recognized, specific inhibition of VEGF, VEGF-receptors, or downstream signaling molecules with the specific intention of inhibiting signaling of this pathway. These agents include but are not limited to: bevacizumab (Avastin™), sorafenib (Nexavar™), sunitinib (Sutent™), axitinib (AG-013736), and AZD 2171.
* Treatment of hypertension with at least 2 or more anti-hypertensive medications with blood pressure remaining greater than 140/90 mmHg.
* Stable management of other toxicities from the cancer treatments
* Expected to continue current cancer treatments for at least 4 weeks
* 18 years and older
* Ability to understand and the willingness to sign a written informed consent document prior to any study specific procedures.

Exclusion Criteria:

* Concurrent use of hematopoietic supportive treatment with erythropoietin or congeners.
* Current uncontrolled toxicities due to the cancer treatments.
* Patients having known contraindications to hydralazine or minoxidil therapy.
* Any readings of systolic blood pressure >200 mmHg or diastolic blood pressure >120 mmHg in the four (4) weeks prior to screening.
* Use of either minoxidil or hydralazine in the six (6) months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydralazine: 25 mg Hydralazine taken twice daily for 1 week, followed by 50 mg taken twice daily for the next week, followed by 100 mg twice daily for the next week
- Minoxidil: 2.5 mg Minoxidil taken twice daily for 1 week, followed by 5 mg taken twice daily for the next week, followed by 10 mg twice daily for the next week
Period: Overall Study
Arm/Group | Hydralazine | Minoxidil
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydralazine | Minoxidil | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 1 | 1
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Change in Blood Pressure
Time Frame: 21 days
Population: No participants analyzed due to poor accrual and insufficient numbers of participants.
Arm/Group | Hydralazine | Minoxidil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Hydralazine | Minoxidil
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydralazine (N=0) | Minoxidil (N=2)
diarrhea (grade 1) (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study enrolled only 2 subjects and due to poor accrual, enrollment was stopped early. Due to the limited number of subjects available results cannot be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No